CLINICAL TRIAL: NCT00470847
Title: A Phase I Study of Lapatinib in Combination With Radiation Therapy in Patients With Brain Metastases From HER2-Positive Breast Cancer
Brief Title: Lapatinib in Combination With Radiation Therapy in Patients With Brain Metastases From HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nancy Lin, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Breast Cancer Research Foundation (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Nancy Lin, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-356
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: Herceptin; breast cancer; radiation therapy; stereotactic radiosurgery; SRS; whole brain radiation; WBRT
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib,Whole Brain Radiation,Herceptin (Other): Lapatinib before and during Whole Brain Radiation Therapy (WBRT), then Herceptin 4mg/kg IV weekly
  Interventions: Drug: Lapatinib; Procedure: Whole Brain Radiation; Drug: Herceptin

INTERVENTIONS:
Drug: Lapatinib — Orally twice daily
  Other Names: Tykerb
Procedure: Whole Brain Radiation — 15 treatments over a period of 3 weeks
Drug: Herceptin — Herceptin 4mg/kg loading dose then 2 mg/kg IV once weekly, then once every three weeks after cycle 3.
  Other Names: Trastuzumab

SUMMARY:
The purpose of this research study is to determine the safety of combining lapatinib plus radiation in patients with breast cancer that has spread to the brain. Depending upon the participants cancer, they may also have stereotactic radiosurgery (SRS). Lapatinib s a compound that may stop cancer cells from growing abnormally. It is thought that lapatinib might also make cancer cells more sensitive to radiation. This drug has been used in other research studies in women with breast cancer, and information from those other research studies suggests that lapatinib may help to shrink or stabilize breast tumors both inside the brain and outside the brain.

DETAILED DESCRIPTION:
* Participant's will be given a study medication-dosing calendar for each treatment cycle. Each treatment cycle lasts four weeks. On the first day of the treatment cycle, participants will take 1 lapatinib orally twice per day, 12 hours apart. After the first day, lapatinib will be taken once a day in the morning.
* Whole brain radiation treatments will begin approximately 1-8 days after the first dose of lapatinib. The radiation treatments will follow standard guidelines and will be supervised by a radiation oncologist. Radiation will be given in 15 treatments over a period of three weeks.
* Some participants will also undergo stereotactic radiosurgery (SRS). SRS is a highly focused and intense form of radiation treatment generally done as an outpatient procedure in a single treatment.
* After whole brain radiation treatments are completed, lapatinib will be continued at the same dose for one more week. After that, the lapatinib dose may change. In addition at the same time, Herceptin will be started. Participants will continue with both lapatinib and herceptin together as long as there is evidence that they are benefitting from it.
* During all treatment cycles participants will have a physical exam and be asked general questions about their health. Photographs will be taken of the tumor, if visible, to assess the response of the tumor to the treatment. An assessment of the tumor by CT scan of the body, and MRI imaging of the brain will be performed every two months. An assessment of heart function by MUGA scan or echocardiogram will be performed every 8 weeks. The participant will also be asked to complete a brief questionnaire measuring quality of life and asking about symptoms related to the cancer at baseline, 6 months, and one year. Blood tests will be performed every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed invasive breast cancer
* HER2 overexpressing breast cancer defined as 3+ staining by immunohistochemistry, or HER2 gene amplification by FISH
* At least one parenchymal brain metastasis
* Disease progression in the CNS as assessed by at least one of the following; new neurological signs or symptoms; new lesion(s) in the CNS on an imaging study; progressive lesions on an imaging study
* At least two weeks since prior radiotherapy, last chemotherapy, immunotherapy, biologic therapy, or major surgery for cancer
* 18 years of age or older
* Life expectancy of greater than 12 weeks
* ECOG performance status 0-2
* Normal organ and marrow function as described in the protocol
* Left ventricular ejection fraction > 50%
* Able to swallow and retain oral medications

Exclusion Criteria:

* Prior WBRT
* Receiving any other investigational agents
* Concurrent chemotherapy, immunotherapy, biologic therapy or hormonal therapy for treatment of their cancer
* History of grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition to herceptin or lapatinib
* Leptomeningeal carcinomatosis as the only site of CNS involvement
* Concurrent treatment with medications that are either inducers of inhibitors of CYP3A4
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or active ulcerative colitis
* History of immediate or delayed hypersensitivity reaction to gadolinium contrast agents
* Other known contraindication to MRI
* Uncontrolled intercurrent illness
* History of other active malignancy except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2007 and December 2009.
Groups:
- Lapatinib,Whole Brain Radiation,Herceptin: Participants received lapatinib, orally, 750mg twice on day one followed by 1000mg, 1250mg, or 1500mg once daily. Whole Brain Radiation therapy (WBRT) (37.5 Gy, 15 fractions) began 1-8 days after starting lapatinib. Lapatinib was continued through WBRT. Following WBRT, patients received trastuzumab intravenously 2mg/kg weekly and lapatinib 1000mg orally once daily.
Period: Overall Study
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Started | 35
Completed | 34
Not Completed | 1
Not completed — Pt still receiving treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 35
Age, Customized [Number; unit: participants]
  Between 30 and 78 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose of Lapatinib When Combined With Cranial Radiation in Patients With CNS Metastases From HER2-positive Breast Cancer.
Description: The maximum tolerated dose is defined as :The highest dose of a drug or treatment that does not cause unacceptable side effects.
Time Frame: 5 Years
Measure: Number; unit: milligrams
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 35
milligrams | 1250

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is the time from date of start of treatment to the date of the first documented progression or death due to any cause. If a patient has not progressed or died, progression free survival is censored at the time of last tumor assessment. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20 % increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 35
months | 4.8 [0 to 58.3]

3. Secondary Outcome: Objective Response Rate in Central Nervous System Sites
Description: Objective Response Rate was defined using volumetric response as the following: Complete Response (CR) is the disappearance of all target lesions, stable/responsive non-target lesions, and no new lesions. Partial response (PR) is at least a 50% reduction in the sum of the target lesions, stable/responsive non-target lesions, and no new lesions. Stable Disease (SD) is neither CR PR or Progressive Disease (PD). And Progressive Disease (PD) is at least 40% increase in sum of target lesionsor the appearance of any new lesion >=6mm in the longest dimension. If a patient progressed in a non-central nervous system(CNS) site first, died, or withdrew from the study for any reason after the first dose of drug was administered, and before a CR or PR in the central nervous system was determined, she was considered a CNS non-responder.
Time Frame: 5 years
Population: 28 participants had measurable disease out of the 35 participants enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 28
percentage of participants | 79 [59 to 92]

4. Secondary Outcome: Percentage of Participants Having Central Nervous System as the Site of the First Progression
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 35
percentage of participants | 23

5. Secondary Outcome: Percentage of Participants Having Non-Central Nervous System Sites as the Site of First Progression
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 35
percentage of participants | 46

6. Secondary Outcome: Overall Survival
Description: Overall average length of participant survival after protocol initiation
Time Frame: Participants were followed for an average of 3.8 years
Measure: Median (Full Range); unit: Months
Arm/Group | Lapatinib,Whole Brain Radiation,Herceptin
Number analyzed (Participants) | 35
Months | 19 [1 to 62]

ADVERSE EVENTS:
Time Frame: May 2007- December 2009
Description: Serious Adverse Events include all Participants N=35. Non-serious Adverse Events also include all participants N=35.
Groups:
- Dose Level 2: n=27 participants Maximum Tolerated Dose 1250 mg lapatinib daily
- Dose Level 1: n=3 participants 1000 mg lapatinib daily
- Dose Level 3: n=5 participants 1500 mg lapatinib daily
Arm/Group | Dose Level 2 | Dose Level 1 | Dose Level 3
Serious Adverse Events (participants affected / at risk) | 8/27 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 27/27 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 2 (N=27) | Dose Level 1 (N=3) | Dose Level 3 (N=5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 2 (N=27) | Dose Level 1 (N=3) | Dose Level 3 (N=5)
Diarrhea (Gastrointestinal disorders) | 21 (21) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (18) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 14 (14) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 0 (0) | 1 (1)
Dehydration (General disorders) | 7 (7) | 0 (0) | 1 (1)
AST/ALT alkaline phosphatase (Hepatobiliary disorders) | 13 (13) | 2 (2) | 3 (3)
Bilirubin (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1)
Anorexia (Gastrointestinal disorders) | 14 (14) | 0 (0) | 2 (2)
Mucositis/chelitis (Infections and infestations) | 5 (5) | 0 (0) | 2 (2)
Ocular (Eye disorders) | 3 (3) | 1 (1) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 9 (9) | 1 (1) | 3 (3)
Lymphocytes/leukocytes (Blood and lymphatic system disorders) | 11 (11) | 2 (2) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2)
Hyperglycemia (Endocrine disorders) | 10 (10) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 8 (8) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 14 (14) | 1 (1) | 2 (2)
Neuropathy-face-motor/taste (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Neuropathy-Sensory (Nervous system disorders) | 7 (7) | 0 (0) | 2 (2)
Neuropathy motor or neurologic-other (Nervous system disorders) | 8 (8) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 4 (4)
Insomnia (General disorders) | 4 (4) | 0 (0) | 2 (2)
Memory Impairment (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 10 (10) | 1 (1) | 2 (2)
Pulmonary/Upper respiratory/cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 3 (3)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 1 (1) | 4 (4)
Rash-Acneiform (Skin and subcutaneous tissue disorders) | 16 (16) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 21 (21) | 3 (3) | 5 (5)
Pain-abdominal (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Pain-back (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Limb, joint, other pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 2 (2)
Kidney function/proteinuria (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No